CLINICAL TRIAL: NCT02454452
Title: Comparative Randomized Clinical Study to Evaluate the Efficacy of Radiofrequency vs Surgical Technique of Internal Saphenous Vein Stripping and CHIVA Technique in the Treatment of Chronic Venous Insufficiency.
Brief Title: Comparison of Radiofrequency, Vein Stripping and CHIVA for Venous Insufficency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Elena González Cañas, MD, PhD, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIC 2012/068
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Varicose Veins
Keywords: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saphenous vein stripping (Active Comparator): Saphenous venous stripping surgical technique
  Interventions: Procedure: Saphenous vein stripping
- CHIVA (Active Comparator): conservative hemodynamic treatment venous insufficiency (CHIVA)
  Interventions: Procedure: CHIVA
- Radiofrequency (Experimental): Radiofrequency treatment applied to the vein with VNUS Closure Fast catheter
  Interventions: Procedure: Radiofrequency

INTERVENTIONS:
Procedure: Radiofrequency — Radiofrequency treatment applied to the vein with VNUS Closure Fast catheter
  Arms: Radiofrequency
Procedure: Saphenous vein stripping — Saphenous vein stripping
  Arms: Saphenous vein stripping
Procedure: CHIVA — conservative hemodynamic treatment venous insufficiency
  Arms: CHIVA

SUMMARY:
Randomized controlled clinical trial aimed to compare the effectiveness and safety of radiofrequency, saphenous vein stripping and conservative hemodynamic treatment of venous insufficiency (CHIVA) in the treatment of saphenous varicose veins, in terms of absence of saphenous vein reflux, patient quality of life and post-surgical complications.

DETAILED DESCRIPTION:
A randomized controlled trial will compare three surgical techniques (stripping, CHIVA and radiofrequency) for the treatment of varicose veins which are currently considered interchangeable standards of care.

The trial will include symptomatic patients with chronic venous insufficiency and saphenous vein insufficiency confirmed by Doppler with diameter greater than 4 mm.

Clinical assessments will be made on first and seventh day after surgery, and then at months 1, 6, 12 and 24. The primary endpoint of the study is the absence of venous reflux in the great saphenous vein segment above-knee. Secondary variables will include VAS for pain and quality of life as assessed by the SF 36 and CIVIQ questionnaires validated in Spanish language. Ultrasound scans will be done the first week and after 1, 6, 12 and 24 months. Intra- and postoperative complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Insufficiency of internal major saphenous vein, confirmed by diameter greater than or equal to 4 mm, assessed by Eco- Dupplex.
* Age > 18 years
* Informed consent

Exclusion Criteria:

* Recurrent varicose veins
* Post-thrombotic syndrome.
* Patients with active malignancies or severe ischemic heart disease.
* Serious liver disease
* Thrombophilia.
* Serious psychiatric diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Absence of venous reflux | 2 years
  Absence of venous reflux by duplex ultrasound

SECONDARY OUTCOMES:
CIVIQ | 2 years
  Venous quality of Life questionnaire - Spanish validated version
SF-36 | 2 years
VCSS | 2 years
  Venous Clinical Severity Score
Surgical complications | 1 month
  Hematoma, echymosis, infection, bleeding, induration, neuritic pain

CONTACTS AND LOCATIONS:
Overall Officials: Elena González Cañas, MD, Principal Investigator — Corporacion Parc Taulí
Locations (1):
- Hospital de Sabadell, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Gonzalez Canas E, Florit Lopez S, Vilagut RV, Guevara-Noriega KA, Santos Espi M, Rios J, Soto SN, Gimenez Gaibar A. A randomized controlled noninferiority trial comparing radiofrequency with stripping and conservative hemodynamic cure for venous insufficiency technique for insufficiency of the great saphenous vein. J Vasc Surg Venous Lymphat Disord. 2021 Jan;9(1):101-112. doi: 10.1016/j.jvsv.2020.04.019. Epub 2020 Apr 28. PMID 32353592